CLINICAL TRIAL: NCT07011836
Title: Enhancing the Effectiveness of Community Health Workers to Reduce Cervical Cancer Disparities in African American Women
Brief Title: Video-Based Patient Navigation to Support Cervical Cancer Screening Among Black Women
Acronym: mNav
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ISA Associates, Inc. (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MD015221; 5R44MD015221-04 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Early Detection of Cancer; Health Behavior; Patient Navigation; African Americans
MeSH Terms: conditions — Uterine Cervical Neoplasms; Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants use an interactive, personalized video-based navigation tool (mNav) and receive navigator support.
  Interventions: Behavioral: mNav Interactive Video + Navigator
- Education Control Group (Active Comparator): Participants view a general cervical cancer education video made for Black women, without personalized content or navigator support.
  Interventions: Behavioral: Educational Video

INTERVENTIONS:
Behavioral: mNav Interactive Video + Navigator — A personalized, video-based tool paired with navigator support to address individual screening barriers.
  Arms: Intervention Group
Behavioral: Educational Video — A culturally tailored cervical cancer education video without additional support or tailoring.
  Arms: Education Control Group

SUMMARY:
The goal of this clinical trial is to test whether an interactive, video-based patient navigation program can improve cervical cancer screening among African American women who are currently overdue for screening.

The main questions it aims to answer are:

Can an interactive video navigation tool (mNav), when paired with in-person navigation, improve screening adherence compared to a standard educational video alone?

Does the intervention improve knowledge, reduce barriers, and increase intentions to get screened?

Researchers will compare participants who receive both the interactive video (guided by an on-screen navigator) and in-person navigation to those who receive only a standard educational video to see if the tailored support increases screening rates.

Participants will:

Complete two phone surveys (one at the beginning and one six months later)

Be randomly assigned to one of two groups:

One group will receive an interactive video experience tailored to their concerns plus support from an in-person navigator

The other group will receive a standard educational video designed for African American women

Have their clinic records reviewed six months later to check for cervical cancer screening completion

ELIGIBILITY:
Inclusion Criteria:

* Black or African American woman
* Nonadherent to USPSTF cervical cancer screening guidelines (no Pap test in the past 3 years or no HPV test in the past 5 years)
* Age 21 to 65 years old
* Not currently pregnant
* No history of hysterectomy
* Access to a mobile phone capable of receiving text messages and watching video content

Exclusion Criteria:

*None

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with a cervix.
Enrollment: 288 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Completion of Cervical Cancer Screening | Within 6 months of enrollment
  Whether participants completed cervical cancer screening, as verified through medical record review. Screening includes a Pap test, HPV test, or co-test, consistent with current guidelines.

SECONDARY OUTCOMES:
Cervical Cancer Screening Intention | Baseline and 6-month follow-up
  Measures participants' self-reported likelihood of obtaining cervical cancer screening in the next 6 months. This is a single-item Likert scale ranging from 0 to 4, with higher scores indicating a greater likelihood of screening. Scale anchors are: 0 = Not at all likely, 1 = A little likely, 2 = Somewhat likely, 3 = Likely, 4 = Very likely.
Cervical Cancer Knowledge Scale | Baseline and 6-month follow-up
  Assessed using a structured survey at baseline and follow-up, this 20-item True/False scale evaluates participant knowledge of cervical cancer risks, screening methods, and guidelines. Scale scores range from 0 to 20, with higher scores indicating greater knowledge. Each correct response is scored as 1; incorrect or missing responses are scored as 0. The total score represents the number of correct responses.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Family and Medical Counseling Service, Inc., Washington D.C., District of Columbia
  - ISA Associates, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The mode of dissemination of public datasets will be via archive files accessible in the public domain. Public datasets will be de-identified so that data cannot be linked to individual research participants
Supporting Information: Study Protocol, ICF
Time Frame: Datasets will be available at a minimum once the data have been accepted for peer-reviewed publication, and earlier if the data are deemed by the PI to be clean and the sharing of data is not expected to inhibit future opportunities for publication.
Access Criteria: A data sharing agreement must be completed and signed by the requesting investigator and the Principal Investigator before this transfer of data can be made.